CLINICAL TRIAL: NCT00539123
Title: Drug Counseling and Abstinent-Contingent Take-Home Buprenorphine in Malaysia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 0506000082; R01DA014718-05A1 (NIH)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Opiate Dependence
Keywords: buprenorphine; drug counseling; HIV risk reduction counseling
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: 2x2 factorial design
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NCB (Experimental): Participants receive Physician Management (PM) and non-contingent provision of take-home doses of buprenorphine-naloxone (NCB).
  Interventions: Behavioral: behavioral drug and HIV risk reduction counseling (BDRC)
- ACB (Experimental): Participants receive Physician Management (PM) and abstinence-contingent provision of take-home doses of buprenorphine-naloxone (ACB).
  Interventions: Behavioral: abstinence-contingent buprenorphine (ACB)

INTERVENTIONS:
Behavioral: behavioral drug and HIV risk reduction counseling (BDRC) — BDRC utilizes short-term behavioral contracts to promote abstinence and reduce drug- and sex-related HIV risk behaviors and can be provided by nurses and medical assistants available in medical settings in Malaysia.
  Arms: NCB
Behavioral: abstinence-contingent buprenorphine (ACB) — Participants achieving heroin abstinence documented by an opioid-negative urine test receive take-home doses of buprenorphine-naloxone, with the number of take-home doses permitted increasing depending on the number of consecutive opioid-negative urine tests. Participants who test positive receive all doses of buprenorphine-naloxone under direct observation in the clinic, using a three-times per week dosing protocol.
  Arms: ACB

SUMMARY:
A randomized clinical trial evaluating whether Behavioral Drug and HIV Risk Reduction Counseling (BDRC), abstinence-contingent take-home buprenorphine (ACB), or the combination of the two improve efficacy and cost-effectiveness of standard buprenorphine treatment for opiate-dependent individuals in Malaysia.

DETAILED DESCRIPTION:
Heroin and injection drug use (IDU) are highly prevalent and driving the HIV epidemic in Malaysia and other countries in the region. In our original RCT, buprenorphine was superior to naltrexone and placebo in treatment retention, weeks of consecutive abstinence and time to heroin use. However, there is room for improvement, since only 50% of subjects assigned to buprenorphine and counseling remained in treatment for 6 months; only 28% avoided relapse to heroin; and treatment reduced drug- but not sex-related HIV risk behaviors. In actual clinical practice in Malaysia and the U.S. buprenorphine treatment effectiveness may be even less, because buprenorphine is provided with relatively minimal psychosocial services (often brief physician management (PM) alone, without additional counseling), and without additional behavioral interventions or contingency management. Hence, we propose a follow up study to evaluate whether standard buprenorphine treatment (consisting of buprenorphine provision, PM, and non-contingent provision of take-home doses of buprenorphine, NCB) is sufficient or whether one or a combination of two behavioral treatments--behavioral drug and HIV risk reduction counseling (BDRC) or abstinence-contingent take-home buprenorphine (ACB)-improve its efficacy. BDRC utilizes short-term behavioral contracts to promote abstinence and reduce drug- and sex-related HIV risk behaviors and can be provided by nurses and medical assistants available in medical settings in Malaysia. ACB, a low cost and feasible alternative to non-contingent take-home buprenorphine (NCB), retains many of its advantages--abstinent patients manage their medication supplies outside of the clinic--but ACB also provides positive incentives for abstinence and directly observed buprenorphine for those with continuing heroin use. In the proposed 2X2 study, heroin dependent patients (N=240) will be inducted onto buprenorphine (weeks 1-2) and then randomized to PM with NCB, PM with ACB, PM with BDRC and NCB, or PM with BDRC and ACB (weeks 3-26). Primary outcome measures include reductions in heroin use (percent days abstinent, proportion of opiate-negative urine tests) and reductions in drug- and sex-related HIV risk behaviors. Data analyses will focus on the intention-to treat sample. The study results will inform practice guidelines and policies regarding buprenorphine treatment.

ELIGIBILITY:
Inclusion Criteria:

* opioid dependence

Exclusion Criteria:

* current dependence on alcohol, benzodiazepines or sedatives current suicide or homicide risk current psychotic disorder or major depression inability to understand protocol or assessment questions life threatening or unstable medical problems more than 3x normal liver enzymes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
reductions in heroin use | 26 weeks
reductions in drug- and sex-related HIV risk | 26 weeks

SECONDARY OUTCOMES:
retention | 26 weeks
reductions in other illicit drug use | 26 weeks
changes in functional status | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Richard S. Schottenfeld, MD, Principal Investigator — Yale University; Mahmud Mazlan, MD, Study Director — Substance Abuse Research Center, Muar
Locations (2):
- Yale University School of Medicine, New Haven, Connecticut, United States
- Substance Abuse Research Center, Muar town, Johor, Malaysia